CLINICAL TRIAL: NCT03148574
Title: Intrauterine Misoprostol Versus Intravenous Oxytocin Infusion During Cesarean Delivery to Reduce Intraoperative and Postoperative Blood Loss: A Randomized Clinical Trial.
Brief Title: Intrauterine Misoprostol Versus Intravenous Oxytocin Infusion During Cesarean Delivery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IUM
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Post Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- misoprostol (Experimental): intrauterine 400 microgram
  Interventions: Drug: Misoprostol
- oxytocin (Active Comparator): intravenous infusion 10 units
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Misoprostol — intrauterine tablets
  Arms: misoprostol
Drug: Oxytocin — intravenous
  Arms: oxytocin

SUMMARY:
Bleeding is still the major cause of mortality and morbidity in postpartum period. World health organization has reported 585000 deaths for pregnancy each year. Twenty five percent of cases die from post-partum bleeding. Mean amount of blood lost is 500 ml during normal vaginal delivery, 1000 ml in cesarean section, and 3500 ml during cesarean section with emergency hysterectomy

ELIGIBILITY:
Inclusion Criteria:

1-Uncomplicated pregnancy, 2-Had no hypersensitivity or contraindications to prostaglandins.

3-Had no history of coagulopathy. 4-Accepting to participate in the study.

Exclusion Criteria:

\1-women with anemia (Haemoglobin <8 gram ). 2 placental abnormality (e.g placenta previa,placenta abruption ) 3. History of complications at previous pregnancy especially postpartum hemorrhage. 4- Maternal hypertension , current or previous history of heart disease ,liver ,Renal disorders or known coagulopathy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-07-02 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
amount of intraoperative blood loss | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No